CLINICAL TRIAL: NCT05431322
Title: Impact of Dexmedetomidine as an Opioid-Sparing Strategy in Thoracoscopic Surgery: A Randomised Controlled Trial
Brief Title: Dexmedetomidine in Thoracoscopic Surgery: Opioid-Sparing Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Kai Wei Hsieh, Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH22-CT2-20
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use; Postoperative Pain
Keywords: Dexmedetomidine; Opioid-free anesthesia; Non-small Cell Lung Cancer
MeSH Terms: conditions — Pain, Postoperative; Carcinoma, Non-Small-Cell Lung | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia (TIVA) + Dexmedetomidine (Experimental): Total intravenous anesthetic drug is propofol. Dexmedetomidine is infused continuously.
  Interventions: Drug: Dexmedetomidine
- Total intravenous anesthesia (TIVA) (No Intervention): Total intravenous anesthetic drug is propofol. The ordinary pain is controlled mainly by opioids.

INTERVENTIONS:
Drug: Dexmedetomidine — Initially give loading dose with 0.5 mcg/kg for 10 min and then keep maintenance dose with 0.5 mcg/kg/h until two-lung ventilation.
  Arms: Total intravenous anesthesia (TIVA) + Dexmedetomidine

SUMMARY:
Numerous studies in recent years have shown that the use of opioid-free analgesia can reduce opioid use and length of stay in the recovery room, as published in the journals Anesthesia & Analgesia1. Compared with traditional opioid analgesic anesthesia, opioid-free analgesic anesthesia can be used to reduce postoperative respiratory complications, postoperative nausea and vomiting, and postoperative opioid needs. During surgery, opioid analgesics may have immunosuppressive effects, but different anesthesia/analgesia methods will change the individual's stress response, affect the human body's cellular immunity, and may even lead to changes in angiogenesis growth factors associated with cancer recurrence, so it is likely to affect the prognosis of cancer patients. In addition, Dexmedetomidine, a highly selective alpha-2 adrenergic receptor agonist, can replace opioids for pain relief during surgery, providing superior analgesia and reducing opioid use while reducing the need for general anesthetics amount, thus avoiding suppression of immune system function. A study in the Journal of Anaesthesiology Clinical Pharmacology pointed out that Dexmedetomidine can be used to replace opioid analgesics in surgical anesthesia, and there was no difference in the use of rescue opioid analgesics during and after surgery5. Several clinical studies have shown that opioid-free anesthesia is significantly associated with a lower incidence of respiratory complications and postoperative nausea and vomiting. Therefore, general anesthesia combined with Dexmedetomidine can be regarded as an opioid-free anesthesia strategy.

DETAILED DESCRIPTION:
Study protocol

All patients received target-controlled infusion (TCI) propofol (3-5 μg ml-1), 2% lidocaine 1.5 mg kg-1 and cisatracurium (0.15-0.2 mg kg-1) or rocuronium (0.6-1.0 mg kg-1).

During induction, the dexmedetomidine group received a loading dose of 0.5 µg kg-1 of dexmedetomidine for 10 minutes. Meanwhile, propofol TCI was started with target of bispectral index set between 40 and 60. After the loading dose was complete, tracheal intubation was performed without opioid analgesic. The following maintenance dose was set as 0.5 µg kg-1 h-1 until the specimen was excised and two-lung ventilation was performed. Dexmedetomidine was then stopped. In contrast, the conventional control group was administered an intermittent bolus dose of fentanyl (0.3-0.5 µg kg-1) to reduce stimuli before tracheal intubation.

In the maintenance phase, parecoxib (40 mg) or propacetamol (1 g) was given if indicated. Anaesthesia was maintained with TCI propofol, and the depth of anaesthesia was monitored using a bispectral index between 40 and 60. Fentanyl was used as a rescue analgesic during the operation. In both groups, when the patient's HR or mean arterial pressure (MAP) was >25% of the baseline, an intermittent bolus dose of 15-25 µg fentanyl was administered. At the end of surgery, patients received intercostal nerve block under thoracoscopy by surgeon.

Haemodynamic stabilisation was achieved in the following situations. If analgesic was administered but the MAP remained elevated at >25% of baseline, nicardipine was considered. If hypotension with MAP dropped >25% from baseline, ephedrine was considered. If bradycardia with HR dropped to <50, atropine was considered.

Pain intensity was assessed in the post-anaesthesia care unit (PACU) using a numerical rating scale (NRS) ranging from 0 to 10 every 15 minutes until 1 hour after surgery. The goal NRS score was <3. If the severity was higher than 3, an intermittent bolus of fentanyl was used. Furthermore, we recorded postoperative complications including nausea, vomiting and respiratory compromise. On the following day, we visited the patient to record complications, severity of postoperative pain and analgesia use in the general ward.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 20 years old and younger than 75 years old
* Diagnosed as stage I-III non-small cell lung cancer
* Received video-assisted thoracoscopic lung wedge resection or lobectomy

Exclusion Criteria:

* Cardiac arrhythmia , such as sinus bradycardia, sinus tachycardia, or high-degree atrioventricular block
* Diagnosed acute myocardial myocardial infarction, congestive heart failure, or stroke within one year
* Patient have underwent coronary artery bypass graft
* Allergy to drug such as Propofol, Sevoflurane, Dexmedetomidine, NSAID, Lidocaine)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The difference in the perioperative dosage of fentanyl between the two groups. | up to post operation day one
  The difference in the perioperative dosage of fentanyl between the two groups.

SECONDARY OUTCOMES:
Postoperative pain scale | up to post operation day one
  The pain scale will be assessed postoperatively
Perioperative hemodynamic parameters | up to post operation day one
  Perioperative blood pressure and heart rate
Postoperative complications | up to post operation day one
  Assessment of nausea and vomiting and respiratory compromise)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan